CLINICAL TRIAL: NCT06468553
Title: Impact of a Multidisciplinary Care Program for Lifestyle Change for Metabolic Control and Quality of Life in Prediabetes: Prediabetes Care Program of Mexico City
Brief Title: Multidisciplinary Care for Lifestyle Change for Metabolic Control and Quality of Life in Prediabetes (PreCPro)
Acronym: PreCPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Especializada en el Manejo de la Diabetes en la Ciudad de Mexico (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101 - 010 - 022 - 23
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: PreDiabetes
Keywords: glycemic control; weight loss; Healthy Lifestyle; Prediabetic State; quality of life; Glucose Metabolism Disorders; Behavior and Behavior Mechanisms; Exercise; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Prediabetic State; Weight Loss; Glucose Metabolism Disorders; Behavior; Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The impact of the intervention on the change in weight and glycated hemoglobin will be determined, secondarily the change in quality of life will also be measured, using a "before and after" design. Subjects who attend the Specialized Diabetes Management Clinic and meet the selection criteria will be included in this study. Once their admission to the study has been decided, subjects will be able to participate in the recruitment and intervention stage and then in the annual follow-up stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prediabetes Care Program (Experimental): Intervention composed of an interdisciplinary care team, patient-centered care approach for behavior change for the adoption of healthy eating and physical activity
  Interventions: Behavioral: Prediabetes Care Program

INTERVENTIONS:
Behavioral: Prediabetes Care Program — Patients are cared for by the medical, nutritionist and psychology team, in a total of 14 individual and group visits, during 12 months of care. The intervention has an initial stage lasting 6 months in which 12 visits will be scheduled and a transition stage lasting 6 more months in which 2 more visits will be scheduled. Patients will be evaluated at 6 months, 12 months and 24 months
  Other Names: PreCPro

SUMMARY:
Prediabetes is part of the natural history of type 2 diabetes mellitus, which is one of the main causes of morbidity and mortality in Mexico. It is known that overweight and obesity are the main risk factors for producing insulin resistance and this in turn leads to prediabetes-diabetes mellitus 2, acting alone or together, excess adipose tissue, mainly visceral, and Prediabetes increase cardiovascular risk before hyperglycemia occurs in the diagnostic criteria for diabetes. Effective strategies have been developed focused on changing lifestyle habits (changes in dietary patterns and increased physical activity) to promote weight loss in populations with and without glucose alterations present, but with limitations in the scope for the size of the affected population. There is a small number of studies developed for this purpose, focused on a multidisciplinary intervention in low- and middle-income countries. The prediabetes care program (PreCPro) is a care initiative developed by the primary care public health services of the Government of Mexico City (CDMX) to promote weight reduction and reduction of hyperglycemia through a intervention composed of an interdisciplinary care team, centered on the patient with a focus on promoting change in people's behavior to adopt healthy eating and physical activity habits. The target population of the prediabetes care program (PreCPro) is made up of patients with prediabetes, without advanced diseases, who receive regular care in public primary care services in Mexico City.

DETAILED DESCRIPTION:
Prediabetes is part of a continuum of progressive dysglycemia that is identified with the presence of hyperglycemia resulting from the destruction or dysfunction of β cells that progresses until plasma glucose concentrations are in the range of diabetes mellitus, by which time the condition has already been detected. presence of organ damage that can no longer be fully reversed and subsequently results in increased disability, morbidity and mortality for families and the high cost of treatment for national healthcare systems. The treatment established for the prevention of diabetes mellitus 2 from stages identifiable through the diagnosis of prediabetes focuses on promoting behavioral changes for the adoption of a healthy diet and increased physical activity with the aim of producing weight reduction with consequent remission of the hyperglycemic state. Although effective behavioral programs have been created for this purpose, the best known being the Diabetes Prevention Program (DPP) in the United States and which is part of its national care strategy, similar care has been carried out in low- and middle-income countries with limited scope because it only focuses on small research studies. The barriers to the implementation of this type of care programs are usually lack of financial resources on the part of health institutions, difficulty in adapting established programs to the specific sociocultural characteristics of each population, lack of access to these programs either due to lack of of time or difficulties in attending due to distance on the part of the participants, among others. Weight loss through changes in dietary patterns and increased physical activity has been shown to prevent or delay the progression of prediabetes to diabetes mellitus 2. The PreCPro program is a care initiative developed by the public health services of primary care of the Government of Mexico City based on the pillars (diet and physical activity) recommended by national and international diabetes mellitus prevention guidelines. The target population of the PreCPro program is made up of patients with prediabetes without advanced diseases, who receive regular care in public primary care services in Mexico City.

ELIGIBILITY:
Inclusion Criteria:

* Having diagnosis of prediabetes
* Acceptance for participation in the program by signing informed consent sheet

Exclusion Criteria:

* Any type of diabetes
* Advanced diseases such as ischemic heart disease, heart failure, KDOQI renal failure ≥1, cerebral vascular disease with functional sequelae or those who have comorbidities that limit their life expectancy such as malignant tumors in advanced stages
* Dependence of illicit drugs
* Conditions that require short-term surgical treatment.
* Pregnancy
* Advanced cognitive deficit or serious psychiatric disorders that hinder treatment adherence
* Use of medications whose use is associated with alterations in blood glucose levels or weight gain or loss, e.g. e.g. metformin, Glucagon-like peptide-1 receptor agonists, orlistat or corticosteroids
* Actively taking any supplements dietary or under naturopathic, homeopathic or alternative therapies
* Have any type of bariatric surgery procedure or weight loss device
* Current participation in another lifestyle, behavior change, or weight loss or gain program or research study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control after the initial stage of the program | six months
  HbA1c (percentage): HbA1c will be compared from the first visit with the visit six months later
Change in weight after the initial stage of the program | six months
  Weight in kilograms. Weight will be compared from the first visit with the visit to six months later

SECONDARY OUTCOMES:
Glycemic control | twenty four months
  HbA1c (percentage): HbA1c will be compared from the last visit (twelve months) and the 24-month visit
Weight change | twenty four months
  Weight change (kg) will be compared from the last visit (twelve months) and the 24-month visit
Lipid control | twenty four months
  Total Cholesterol, HDL-Cholesterol, Non-HDL Cholesterol and triglycerides in mg/dL will be compared from the last visit (twelve months) and the 24-month visit
Blood pressure | twenty four months
  Systolic and diastolic blood pressure (mmHg) will be compared from the last visit (twelve months) and the 24-month visit
Health-related Quality of Life perception assessed by EuroQol (EQ-5D) Visual Analogue Scale questionnaire | twenty four months
  Health-related Quality of life perception with EQ-5D questionnaire visual analogue scale (0-100, higher score means better self-care). Health-related Quality of Life will be compared from the last visit (twelve months) and the 24-month visit
Glycemic control | twelve months
  HbA1c (percentage): HbA1c will be compared from the visit on the six months with the last visit (12 month)
Weight change | twelve months
  Weight Change in kilograms will be compared from the visit on the six months with the last visit (12 month)
Lipid control | twelve months
  Total Cholesterol, HDL-Cholesterol, Non-HDL Cholesterol and triglycerides in mg/dL will be compared from the visit on the six months with the last visit (12 month)
Blood pressure | twelve months
  Systolic and diastolic blood pressure (mmHg) will be compared from the visit on the six months with the last visit (12 month)
Health-related Quality of Life perception assessed by EuroQol (EQ-5D) Visual Analogue Scale questionnaire | twelve months
  Health-related Quality of life perception with EQ-5D questionnaire visual analogue scale (0-100, higher score means better self-care). Health-related Quality of Life will be compared from the visit on the six months with the last visit (12 month)
Lipid control | six months
  Total Cholesterol, HDL-Cholesterol, Non-HDL Cholesterol and triglycerides in mg/dL will be compared from the first visit with the visit to six months late
Blood pressure | six months
  Systolic and diastolic blood pressure (mmHg) will be compared from the first visit with the visit to six months later
Health-related Quality of Life perception assessed by EuroQol (EQ-5D) Visual Analogue Scale questionnaire | six months
  Health-related Quality of life perception with EQ-5D questionnaire visual analogue scale (0-100, higher score means better self-care). Health-related Quality of Life will be compared from the first visit with the visit to six months later

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Silva-Tinoco, MD, Study Director — Clinica Especializada en el Manejo de la Diabetes; Viridiana De la Torre-Saldaña, MD, Principal Investigator — Clinica Especializada en el Manejo de la Diabetes
Locations (1):
- Clinica Especializada en el Manejo de la Diabetes, Mexico City, Iztapalapa, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The availability to share any data from individual participants must be requested primarily to the institutional Research and Ethics Committee by the study investigators.

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF DIABETES ATLAS [Internet]. 10th edition. Brussels: International Diabetes Federation; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK581934/ PMID 35914061
- [Background] Basto-Abreu A, Lopez-Olmedo N, Rojas-Martinez R, Aguilar-Salinas CA, Moreno-Banda GL, Carnalla M, Rivera JA, Romero-Martinez M, Barquera S, Barrientos-Gutierrez T. Prevalencia de prediabetes y diabetes en Mexico: Ensanut 2022. Salud Publica Mex. 2023 Jun 13;65:s163-s168. doi: 10.21149/14832. Spanish. PMID 38060942